CLINICAL TRIAL: NCT05240846
Title: Paramedian Approach for Spinal Anesthesia Using Ultrasound Assistance Versus Conventional Palpation in Morbidly Obese Patients: A Randomized Controlled Trial
Brief Title: Spinal Anesthesia Using Ultrasound Assistance Versus Conventional Palpation in Morbidly Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed Fouad Algyar, Doctor, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MKSU 48-1-31
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Spinal Anesthesia; Ultrasound Assistance; Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paramedian conventional palpation group (Experimental): Patients in this group underwent conventional landmark guided paramedian spinal anesthetic. The spinal anesthesia will be administered based on conventional landmark-based paramedian approach.
  Interventions: Procedure: Paramedian conventional palpation group
- Ultrasound assistance paramedian spinal group (Experimental): This group will have their spinal anesthetic done based on Ultrasound assistance paramedian spinal.
  Interventions: Procedure: Ultrasound assistance paramedian spinal group

INTERVENTIONS:
Procedure: Paramedian conventional palpation group — Patients in this group underwent conventional landmark guided paramedian spinal anesthetic. The spinal anesthesia will be administered based on conventional landmark-based paramedian approach.
  Arms: Paramedian conventional palpation group
Procedure: Ultrasound assistance paramedian spinal group — This group will have their spinal anesthetic done based on ultrasound assistance paramedian spinal. Spinal anesthesia with a paramedian approach was performed based on the optimum puncture point, suggested puncture angles, and puncture depth. The suggested puncture angles included the cephalad angle measured by the built-in angle program of the ultrasound and the medial angle measured by a 180° protractor (Deli). The puncture depth, the distance from the skin to the posterior complex, was measured utilizing the ultrasound clipper tool.
  Arms: Ultrasound assistance paramedian spinal group

SUMMARY:
The aim of this study is to compare the paramedian approach for spinal anesthesia using ultrasound assistance (USAS) versus conventional palpation in morbidly obese patients undergoing elective surgeries.

DETAILED DESCRIPTION:
Performing spinal anesthesia using a conventional approach can be considerably challenging in obese patients. Multiple needle attempts may lead to a higher incidence of complications (e.g., postdural puncture headache, paresthesia, hematoma, and infection) and increase patient discomfort and dissatisfaction. Therefore, novel techniques are needed to improve the success rate of spinal anesthesia for such patients.

There are two puncture approaches for spinal anesthesia: median approach puncture and paramedian approach puncture. Early studies have noted that the success rate of paramedian approach puncture was higher than that of median approach puncture and that it is associated with fewer complications and postoperative complications.

A paramedian approach has been shown to improve the success rate of spinal anesthesia, especially in patients who are unable to sit up or those with a degenerative spine condition. The use of ultrasound has been suggested to increase the efficacy of spinal anesthesia.

Recently, ultrasound has emerged as a way to facilitate lumbar neuraxial blocks, namely, the ultrasound assistance (USAS) technique. The ultrasound assistance technique is beneficial for lumbar neuraxial anesthesia, improving technique performance by providing reliable anatomical information.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both sexes
* Body mass index (BMI) ≥ 40 kg/m2
* Patients undergoing elective surgeries

Exclusion Criteria:

* Rejection of spinal anesthesia
* History of spinal deformity or spinal surgery
* Contraindications to spinal anesthesia (infection of the puncture site, coagulation dysfunction, allergy to local anesthesia, insufficient blood volume or abnormal spinal anatomy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
The rate of successful dural puncture on the first attempt | Intraoperatively
  First-attempt success rate will be recorded

SECONDARY OUTCOMES:
Total success rate of spinal anesthesia | Intraoperatively
  Successful Dural Puncture Rates for Selected Number of Attempts and Passes in both intervention groups
Adverse reactions during puncture | Intraoperatively
  Adverse reactions during puncture as incidence of nerve stimulation
Complications after anesthesia | 24 hours Postoperative
  Complications after anesthesia as incidence of low back pain
Patients' satisfaction after surgery | 24 hours Postoperative
  6- Degree of patient satisfaction will be assessed on a 3-point scale; (1= unsatisfied 2= neither satisfied nor unsatisfied 3= satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Kafr El-Sheikh University Hospitals, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
This study will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study